CLINICAL TRIAL: NCT05294536
Title: A Randomized, Open-label, Two-period, and Double-cross Comparative Study on the Pharmacokinetics of Liraglutide Injection (RD12014) and Victoza® in Healthy Volunteers
Brief Title: A Pharmacokinetic Study Comparing the Liraglutide Injection (RD12014) and Victoza® in Healthy Chinese Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sunshine Lake Pharma Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 12014-P-01/CRC-C1944
Record Dates: First submitted 2022-03-10; First posted 2022-03-24 (Actual); Last update posted 2022-03-24 (Actual); Status verified 2022-03

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Liraglutide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Liraglutide injection (RD12014)+ Victoza (Experimental): Subjects receive liraglutide injection(RD12014) in the first cycle and Victoza in the second cycle.
  Interventions: Drug: Liraglutide injection,RD12014; Drug: Liraglutide injection,Victoza
- Victoza + Liraglutide injection (RD12014) (Experimental): Subjects receive Victoza in the first cycle and liraglutide injection(RD12014) in the second cycle.
  Interventions: Drug: Liraglutide injection,RD12014; Drug: Liraglutide injection,Victoza

INTERVENTIONS:
Drug: Liraglutide injection,RD12014 — single dose, s.c. injection
Drug: Liraglutide injection,Victoza — single dose, s.c. injection

SUMMARY:
To evaluate the pharmacokinetics similarity between the liraglutide injection (RD12014) produced by Sunshine Lake Pharma Co., Ltd. and liraglutide injection (Victoza®) produced by Novo Nordisk Pharmaceutical Co., Ltd for single dose in healthy male subjects, as well as to evaluate the similarity of the safety and immunogenicity between RD12014 and Victoza ® in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* 1. Being willing to participate in the experiment, fully understand and sign the informed consent, fully understand and able to complete the experiment according to the requirements of the experiment protocol;
* 2. Aged between 18 and 45 years old of healthy male subjects ;
* 3. Weight ≥50kg, and body mass index(BMI)= 19.0-26.0 kg/m2 ;
* 4. No history of respiratory system, cardiovascular system, digestive system, urinary system, hematological system, endocrine system,nervous system or metabolic abnormalities;
* 5. Normal or abnormal vital signs, physical examination, laboratory examination, electrocardiogram, abdominal ultrasound examination and chest X-ray examination have no clinical significance;

Exclusion Criteria:

* 1. Have a history of fainting needles, fainting blood;
* 2. Positive for hepatitis (including hepatitis B and C), HIV or syphilis at screening;
* 3. Have taken any prescription, over-the-counter, herbal medicine or health care products (other than normal vitamin products)within 2 weeks prior to the use of the study drug;
* 4. Have a history of taken Liraglutide or other human glucagon-like peptides-1 analogues before the trial;
* 5. Those who have been screened positive for drugs at screening;
* 6. Donated blood (> 400 ml) within 3 months before taking the study drug;
* 7. Heavy smoker or those who smoked more than 10 cigarettes per day before taking the study drug.
* 8. Alcohol abuse (drinking 21 units of alcohol per week: 1 unit = 360 ml of beer or 45 ml of 40% alcoholic spirits or 150 ml of wine) or positive for breath alcohol test ;
* 9. Those who have been screened positive for drugs or have a history of drug abuse;
* 10. Known allergy to Liraglutide or any of the excipients of the formulation;
* 11. Those who have a history or family history of medullary thyroid cancer (grandparents, parents and siblings), or inherited diseases that predispose them to medullary thyroid cancer;Or have a history or family history of multiple endocrine adenomatosis;
* 12. Have participated in the drug clinical trial and taken the test drug within 3 months before taking the study drug;
* 13. During the trial period and within 3 months after the last dose, those who want their female partners to become pregnant or is unwilling to use reliable contraceptive methods
* 14. Other cases judged by researchers to be unsuitable for selection.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2020-06-22 (Actual); Primary Completion 2020-07-20 (Actual); Study Completion 2020-11-27 (Actual)

PRIMARY OUTCOMES:
Maximum (peak) plasma drug concentration(Cmax) | 0 hour（pre-dose,within 30mins） to 72 hours after administration
  Maximum (peak) plasma drug concentration
Area under the plasma concentration-time curve from time zero to time t (AUC0-t) | 0 hour（pre-dose,within 30mins） to 72 hours after administration
  The area under the plasma concentration curve from 0 to 72 h

SECONDARY OUTCOMES:
Area under the plasma concentration-time curve from time zero to ∞ (AUC0-∞) | 0 hour（pre-dose,within 30mins） to infinity after administration
  The area under the plasma concentration curve from 0 to ∞
Time to reach maximum plasma concentration following drug administration (Tmax) | 0 hour（pre-dose,within 30mins） to 72 hours after administration
  Time to maximum concentration
Elimination half-life (t1/2) | 0 hour（pre-dose,within 30mins） to 72 hours after administration
  Elimination half-life
Apparent total body clearance (CL/F) | 0 hour（pre-dose,within 30mins） to 72 hours after administration
  Apparent total body clearance
Apparent volume of distribution (Vd/F) | 0 hour（pre-dose,within 30mins） to 72 hours after administration
  Apparent volume of distribution
Adverse Event, Serious Adverse Event | Up to day 4 after the second dose.
  Monitor the safety indicators of subjects during the trial

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Xuhui Central Hospital, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Derived] Zhou R, Guo L, Gao X, Wang Y, Xu W, Zou Y, Li W, Zhuang Y, Liu G, Liu Y. A phase I study comparing the pharmacokinetics of the biosimilar (RD12014) with liraglutide (Victoza) in healthy Chinese male subjects. Clin Transl Sci. 2022 Oct;15(10):2458-2467. doi: 10.1111/cts.13374. Epub 2022 Jul 31. PMID 35871497